CLINICAL TRIAL: NCT02826317
Title: Evaluation du caractère Neuropathique Des Douleurs Post opératoires. Enquête 2 Jours : DN4-SFAR
Brief Title: Neuropathic Evaluation of Postoperative Pain
Acronym: DN4-SFAR
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 14.02
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Neuropathic Pain Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: preoperative and postoperative setting — Preoperative assessment will consist on collecting demographic data as well as the presence preoperative chronic pain and its localization, preoperative opioid, gabapentin or pregabalin consumption. In postoperative, we will collect the following data: type of anesthesia, intra operative ketamine administration, type and total dose of opioid administered during surgery. Pain will be evaluated at least 2 hours after the surgery within the same day (D0) and then at day 2 (D2), 1 (M1) and 2 months (M2) after the surgery. Pain will be assessed using a 10-point NPS. If NPS >0, neuropathic pain will be diagnosed on the basis of DN4 questionnaire. NCPSP is defined by NPS >0 and positive DN4 (DN4 ≥ 4 /10) (11). APSNP and CPSNP are defined by D0/D2 DN4≥ 4/10 and M1/M2 DN4≥ 4/10, respectively.

SUMMARY:
Chronic postsurgical pain (CPSP) is defined by pain persisting longer than 2 months after surgery (1). Its incidence varies from 10 to 50 % in the literature (2). A high proportion of CPSP is neuropathic (CPSNP) (4). Postoperative pain is traditionally classified as nociceptive pain and the more intense is this pain on a numeric pain scale (NPS), higher are the risks of pain chronicization and the duration of the severe pain is longer (5,6). However, acute neuropathic pain (ANP) can be present in the postoperative setting. However, data on the prevalence of ANP immediately after surgery are scarce and no screening tool has been validated so far in this setting. Therefore, the first objective of this multicenter observational study is to prospectively describe the incidence of APSNP in a large population using the DN4 questionnaire. The second objective of our study is to confirm the hypothetic link between APSNP and CPSNP at 1 and 2 months after surgery in a large population. It is hypothesized that the systematic use of the DN4 questionnaire in postoperative could help detect patients at risk of CPSNP.

DETAILED DESCRIPTION:
Chronic postsurgical pain (CPSP) is defined by pain persisting longer than 2 months after surgery (1). Its incidence varies from 10 to 50 % in the literature (2). A high proportion of CPSP is neuropathic (CPSNP) (4). Postoperative pain is traditionally classified as nociceptive pain and the more intense is this pain on a numeric pain scale (NPS), higher are the risks of pain chronicization and the duration of the severe pain is longer (5,6). However, acute neuropathic pain (ANP) can be present in the postoperative setting. However, data on the prevalence of ANP immediately after surgery are scarce and no screening tool has been validated so far in this setting. Therefore, the first objective of this multicenter observational study is to prospectively describe the incidence of APSNP in a large population using the DN4 questionnaire. The second objective of our study is to confirm the hypothetic link between APSNP and CPSNP at 1 and 2 months after surgery in a large population. It is hypothesized that the systematic use of the DN4 questionnaire in postoperative could help detect patients at risk of CPSNP.

Methods:

Investigators and centers will be recruited through the SFAR (French Society of Anesthesiology and Intensive Care) research network. The study will take place during the same 2 consecutive days in all the centers in France. Each center agreed to include as many patients as they could during this period. All adult patients undergoing inpatient scheduled or urgent surgery are eligible. The study is solely observational and does not interfere with the patient's care. Preoperative assessment will consist on collecting demographic data (age, sex, body mass index, type of surgery) as well as the presence preoperative chronic pain and its localization, preoperative opioid, gabapentin or pregabalin consumption. In postoperative, we will collect the following data: type of anesthesia, intra operative ketamine administration, type and total dose of opioid administered during surgery. Pain will be evaluated at least 2 hours after the surgery within the same day (D0) and then at day 2 (D2), 1 (M1) and 2 months (M2) after the surgery. Pain will be assessed using a 10-point NPS. If NPS >0, neuropathic pain will be diagnosed on the basis of DN4 questionnaire. NCPSP is defined by NPS >0 and positive DN4 (DN4 ≥ 4 /10) (11). APSNP and CPSNP are defined by D0/D2 DN4≥ 4/10 and M1/M2 DN4≥ 4/10, respectively. The preoperative and immediate postoperative (day 0 and day 2) data will be collected by one investigator in each center. The latter data (1 and 2 months after the surgery) will be assessed over the phone by research nurses.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing inpatient scheduled or urgent surgery

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing inpatient scheduled or urgent surgery are eligible
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
prospectively describe the incidence of APSNP in a large population using the DN4 questionnaire | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Hélène BELOEIL, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beloeil H, Sion B, Rousseau C, Albaladejo P, Raux M, Aubrun F, Martinez V; SFAR research network. Early postoperative neuropathic pain assessed by the DN4 score predicts an increased risk of persistent postsurgical neuropathic pain. Eur J Anaesthesiol. 2017 Oct;34(10):652-657. doi: 10.1097/EJA.0000000000000634. PMID 28437260